CLINICAL TRIAL: NCT01507558
Title: Dexamethasone Infusion to the Adventitia to Enhance Clinical Efficacy After Femoropopliteal Revascularization
Acronym: DANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Warren J. Gasper, MD, MD, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-02101
Record Dates: First submitted 2011-11-09; First posted 2012-01-11 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Femoral popliteal lesions
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty; Atherectomy; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Perivascular administration of dexamethasone following endovascular superficial femoral and popliteal artery angioplasty or atherectomy.
  Interventions: Procedure: Administration of dexamethasone to SFA/popliteal adventitia

INTERVENTIONS:
Procedure: Administration of dexamethasone to SFA/popliteal adventitia — Following a balloon angioplasty or atherectomy of a stenotic TASC II A, B, or C lesion in the superficial femoral or popliteal artery, a Bullfrog Micro-Infusion Catheter will be used to infuse 0.96 mg dexamethasone per cm arterial lesion.
  Other Names: angioplasty; atherectomy; TASC II A, B, C lesion; dexamethasone; superficial femoral artery; popliteal artery

SUMMARY:
The purpose of this study is to test if dexamethasone, an anti-inflammatory medication approved by the US Food and Drug Administration (FDA), can be injected safely into the tissue around the blood vessel wall at the time of an angioplasty or atherectomy.

DETAILED DESCRIPTION:
This is an investigator-initiated, single-arm, external pilot study to assess the safety and feasibility of perivascular administration of dexamethasone following endovascular superficial femoral and popliteal artery angioplasty or atherectomy.

Although dexamethasone is approved by the FDA for injection into blood, skin or joints, it has not been approved by the FDA for injection around blood vessels. The investigators want to find out if this procedure helps prevent re-narrowing of the blood vessel after angioplasty or atherectomy. The dexamethasone will be injected with a Bullfrog® Micro-Infusion catheter, which is an FDA-approved device for injecting medications into tissues around the blood vessel wall. The Bullfrog® Micro-Infusion catheter is similar to other balloon tipped catheters except that it contains a microneedle covered by a fold of semi-rigid balloon. Once the balloon is inflated, the microneedle is uncovered and a medication can be injected into the tissue around the blood vessel.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 40 years and < 80 years of age
* Patient has severe, lifestyle-limiting claudication or critical limb ischemia (Rutherford classification 3-6)
* Patient has TASC II A, B or C disease, SFA revascularization is preferred over medical management, and endovascular approach is preferred revascularization strategy
* Patient has a resting ABI of <0.9 or an abnormal treadmill ABI. Patients with incompressible arteries must have a TBI <0.8
* Patient has at least 1 infra-popliteal run-off vessel with patency to the ankle without a >50% stenosis
* Successful crossing of the lesion with guidewire and successful atherectomy or angioplasty with residual stenosis <30% as compared to the reference vessels
* Atherectomy procedure does not result in embolization, arteriovenous fistula or perforation
* Patient agrees to return for a clinical assessment duplex ultrasound at 1, 3, 6, 9, 12 and 24 months (routine clinical care)

Exclusion Criteria:

* Patient is simultaneously participating in another investigational drug or device study
* Patient is pregnant or breast-feeding
* Patient has cancer, autoimmune disease, bone marrow or organ transplant, or other concurrent medical illness requiring immunosuppressive therapy
* Patient has end-stage renal disease and chronic kidney disease (eGFR<30)
* Patient has an active infection
* Patient has a known hypersensitivity or contraindication to heparin, contrast agents, excipients of Dexamethasone Sodium Phosphate Injection, USP, dexamethasone, or other glucocorticoids
* Patient has a life expectancy of less than one year

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety Outcome Measures: | 30 days
  Freedom from death, vessel dissection, thrombosis or extravasation at 30 days post-procedure.
Effectiveness Outcome Measures: | 6 months
  Freedom from Target Lesion Revascularization (TLR) and/or Target Vessel Revascularization (TVR) at 6 months post-procedure.

SECONDARY OUTCOMES:
Safety Outcome Measures: | 24 months
  Freedom from death, stroke, myocardial infarction, emergent surgical revascularization, significant distal embolization in target limb, and thrombosis of target vessel

CONTACTS AND LOCATIONS:
Overall Officials: Warren J. Gasper, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco Medical Center, San Francisco, California

REFERENCES:
- [Derived] Owens CD, Gasper WJ, Walker JP, Alley HF, Conte MS, Grenon SM. Safety and feasibility of adjunctive dexamethasone infusion into the adventitia of the femoropopliteal artery following endovascular revascularization. J Vasc Surg. 2014 Apr;59(4):1016-24. doi: 10.1016/j.jvs.2013.10.051. Epub 2014 Jan 11. PMID 24423476